CLINICAL TRIAL: NCT05259488
Title: Preoperative Immunonutrition in Laparoscopic Total D2 Gastrectomy: a Single-centre Comparative Study
Brief Title: Preoperative Immunonutrition in Laparoscopic Total D2 Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Prof, University of Rome Tor Vergata
Other Study IDs: Protocollo xx/22
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer; Surgery; Laparoscopic; Gastric Neoplasm; Digestive Cancer
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients receiving immunonutrition supply: Dietary Supplement: Immunonutrition nutridrinks 3 times a day 5 days prior surgery plus maltodextrins the day of surgery
  Interventions: Dietary Supplement: immunonutrition
- historical control group: standard dietary advice

INTERVENTIONS:
Dietary Supplement: immunonutrition — nutridrinks 3 times a day 5 days prior surgery plus maltodextrins the day of surgery
  Groups: patients receiving immunonutrition supply

SUMMARY:
Immunonutrition (IN) appears to reduce infective complications and in-hospital length of stay (LOS) after gastrointestinal surgery. More specifically, it seems to be beneficial also in gastric cancer surgery. Potential benefits of combining preoperative IN (PIN) with protocols of enhanced recovery after surgery (ERAS) in reducing LOS in laparoscopic total gastrectomy are yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Primary gastric cancer
* Preoperative staging I-III
* Eligible for laparoscopic D2 total gastrectomy

Exclusion Criteria:

* Acquired or congenital immunodeficiency
* Malnutrition (MNA-SF score < 12)
* Preoperative infection
* Previous gastric surgery
* ASA IV
* Emergency setting
* Para-aortic node involvement
* Intraoperative evidence of distant metastasis or peritoneal carcinosis
* Conversion to open surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All normonourished patients undergoing elective ERAS laparoscopic total gastrectomy for cancer at Minimally Invasive Surgery Unit of Tor Vergata University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
30-days postoperative complications | up to 30 days after discharge
  Rate of any complication after colorectal resection
LOS | up to 30 days after discharge
  number of days between primary colorectal resection and discharge

SECONDARY OUTCOMES:
Anastomotic leak | up to 30 days after discharge
  rate of any postoperative leakage of oesophagojejunal, jejunojejunal anastomosis, clinically, radiologically or endoscopically demonstrated
Pneumonia | up to 30 days after discharge
  rate of radiologically demonstrated pneumonia
Ileus | up to 30 days after discharge
  rate of any ileus clinically demonstrated
Prolonged length of stay | up to 30 days after discharge
  rate of any patient discharged after 15 days
Readmission | up to 30 days after discharge
  Rate of any unplanned readmission after discharge
Mortality | up to 30 days after discharge
  Rate of any mortality
Time of first defacation | up to 30 days after discharge
  time to first bowel opened to stool
Time of tolerated fluid intake | up to 30 days after discharge
  time to first tolerated fluid intake
Time of tolerated food intake | up to 30 days after discharge
  time to first tolerated food intake

IPD SHARING:
Plan to Share IPD: No
data available on request

REFERENCES:
- [Derived] Franceschilli M, Siragusa L, Usai V, Dhimolea S, Pirozzi B, Sibio S, Di Carlo S. Immunonutrition reduces complications rate and length of stay after laparoscopic total gastrectomy: a single unit retrospective study. Discov Oncol. 2022 Jul 11;13(1):62. doi: 10.1007/s12672-022-00490-5. PMID 35816241